CLINICAL TRIAL: NCT05934890
Title: A Phase 3, Randomized, Blinded, Active-controlled Study to Evaluate the Immunogenicity and Safety of Walvax's 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV13-TT) as Compared to Pfizer's 13-Valent Pneumococcal Conjugate Vaccine (PCV13) Co-administered With EPI Vaccines at 2, 4, and 12-15 Months of Age, to Healthy Infants in Indonesia
Brief Title: A Phase 3 Study to Evaluate the Immunogenicity and Safety of Walvax's PCV13-TT as Compared to Pfizer's PCV13
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PCV13-004
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pneumococcal Disease, Invasive
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Active-controlled
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walvax PCV13-TT (Experimental): Primary Vaccination: A total of approximately 300 infants 6-8 weeks of age will be enrolled and assigned randomly to receive at 2, 4, and 12-15 months of age 1 dose of PCV13-TT. Standard EPI vaccines will be administered concomitantly.
  Booster Vaccination: At 12-15 months of age (8 to 11 months after the 2nd dose of the primary series), infants will receive a booster dose of PCV13-TT.
  Interventions: Biological: Walvax PCV13-TT
- Pfizer PCV13 (Active Comparator): Primary Vaccination: A total of approximately 300 infants 6-8 weeks of age will be enrolled and assigned randomly to receive at 2, 4, and 12-15 months of age 1 dose of PCV13. Standard EPI vaccines will be administered concomitantly.
  Booster Vaccination: At 12-15 months of age (8 to 11 months after the 2nd dose of the primary series), infants will receive a booster dose of PCV13.
  Interventions: Biological: Pfizer PCV13

INTERVENTIONS:
Biological: Walvax PCV13-TT — PCV13-TT is supplied as 0.5 mL prefill syringe (PFS), with 0.5 mL suspension for intramuscular injection. After shaking, the vaccine is a homogenous, white suspension. Each dose (0.5 mL) of PCV13-TT contains pneumococcal polysaccharide serotypes 1, 3 4, 5, 6A 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F which are conjugated to TT carrier protein individually.
  The vaccine is formulated in phosphate-buffered saline containing 4.25 mg/dose sodium chloride (NaCl), 44.35 μg/dose sodium dihydrogen phosphate (NaH2PO4), 19.0 μg/dose disodium hydrogen phosphate (Na2HPO4), and contains 0.5 mg/dose of aluminum phosphate as an adjuvant; no preservatives added.
  Arms: Walvax PCV13-TT
Biological: Pfizer PCV13 — PCV13 is a suspension for intramuscular injection available in 0.5 mL single-dose prefilled syringes. Each 0.5 mL dose of PCV13 is formulated to contain approximately 2.2 μg of each of S. pneumoniae serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F polysaccharides, 4.4 μg of 6B polysaccharides, 34 μg 26 CRM197 carrier protein, 100 μg polysorbate 80, 295 μg succinate buffer and 125 μg aluminum as aluminum phosphate adjuvant.
  Arms: Pfizer PCV13

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity and safety of a novel 13-valent pneumococcal polysaccharide conjugate vaccine (PCV13-TT) as compared to Pfizer's 13-valent pneumococcal conjugate vaccine (PCV13) when co-administered with local EPI Vaccines at 2, 4, and 12-15 months of age, to healthy infants in Indonesia. This study aims to demonstrate the non-inferiority of the serotype-specific immune responses elicited by the novel PCV13-TT as compared to PCV13 one month after the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Infants must meet ALL the following inclusion criteria for enrollment in the study, at the time of the screening:

  1. Healthy infants based on medical history and clinical assessment.
  2. Age of 6-8 weeks at enrolment. Infants will be eligible since the day they reach 6 weeks of age and until 8 weeks of age included.
  3. Body weight at enrollment ≥3.5 kg.
  4. Infant's parent(s) or legal guardian(s) must be able and willing to provide voluntary written/thumb-printed informed consent for the infant to participate in the study.
  5. Infant's parent(s) or legal guardian(s) must be able to comprehend and comply with study requirements and procedures and must be willing and able to return or make themselves available for all scheduled follow-up visits.
  6. Infant's parents must have a readily identifiable place of residence in the study area, be available for the duration of trial participation, and have means of telephone contact.

Exclusion Criteria:

* The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

  1. Use of any investigational medicinal product prior to randomization or planned use of such a product during the period of study participation.
  2. History of S. pneumoniae infection as confirmed by medical enquiry or as confirmed by laboratory testing if available.
  3. Participant has fever (axillary temperature ≥ 37.5℃) within 24 hours prior to the 1st dose of vaccination; (If the subject does not meet the criteria, the visit may be rescheduled when the criteria are met.)
  4. The infant who are children in care, preterm and low-birth-weight(Preterm infants have a gestational age below 37 weeks at birth and low-birth-weight infants have a birth weight below 2.5 kg).
  5. History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the 2 study vaccines. This includes all components of the EPI vaccines.
  6. History of anaphylactic shock.
  7. Any abnormal vital sign.
  8. Any moderate or severe acute illness.
  9. History of administration of a non-study vaccine within 30 days prior to administration of study vaccine, other than EPI vaccinations (Note: EPI vaccines other than that stipulated in the study must be given at least 14 days prior to the investigational vaccine.)
  10. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for 14 days at a dose of 20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, epidural, or topical (skin or eyes) corticosteroids within indicated dosage are permitted.
  11. Administration of immunoglobulins and/or any blood products or anticipation of such administration during the study period.
  12. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding (e.g., thalassemia, coagulation factor deficiencies, severe anemia at birth).
  13. History of suspected primary immunodeficiency.
  14. History of meningitis, seizures or any neurological disorder.
  15. A family history of congenital or hereditary immunodeficiency.
  16. The infant is a direct descendant (child or grandchild) of any person employed by the Sponsor, the CRO, the investigator, study site personnel.
  17. Any medical or social condition that in the opinion of the investigator may compromise the well-being of the study participant, interfere with the study objectives, pose a risk to the study participant, or prevent the study participant from completing the study follow-up.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 630 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity and non-inferiority as measured by serotype-specific IgG | 1 month after the booster dose
  Percentage of infants with serotype-specific IgG concentrations ≥0.35 μg/mL
Immunogenicity and non-inferiority as measured by serotype-specific IgG GMC | 1 month after the booster dose
  Serotype-specific IgG GMCs

SECONDARY OUTCOMES:
Solicited local and systemic adverse events after each dose | within 30 min and 7 days after each dose
  Frequency and severity of solicited local and systemic adverse events (AEs)
Unsolicited adverse events after each dose | within 30 days after each dose
  Frequency and severity of unsolicited AEs
Serious adverse events throughout the study | from dose 1 until 6 months after booster dose
  Frequency of serious AEs (SAEs)
Immune response to primary series as measured by serotype-specific IgG | 1 month after the 2nd dose
  Percentage of infants with pneumococcal serotype-specific IgG concentrations ≥0.35 µg/mL
Immune response to primary series as measured by serotype-specific IgG GMC | 1 month after the 2nd dose
  Serotype-specific IgG GMCs
Functional antibody responses as measured by serotype-specific OPA titer | baseline, 1 month after the 2nd dose, before the booster dose, and 1 month after the booster dose
  Percentage of infants with serotype-specific OPA titer ≥1:8
Functional antibody responses as measured by serotype-specific OPA geometric mean titers (GMTs) | baseline, 1 month after the 2nd dose, before the booster dose, and 1 month after the booster dose
  Serotype-specific OPA geometric mean titers (GMTs)
Immune persistence as measured by serotype-specific IgG | 12-15 months of age, before the booster dose
  Percentage of infants with pneumococcal serotype-specific IgG concentrations ≥0.35 µg/mL
Immune persistence as measured by serotype-specific IgG GMC | 12-15 months of age, before the booster dose
  Serotype-specific IgG GMCs

OTHER OUTCOMES:
Exploratory_Non-interference | 1 month after the 2nd dose
  Percentage of infants with anti-diphtheria toxoid IgG concentrations ≥0.1 IU/mL
Exploratory_Non-interference | 1 month after the 2nd dose
  Percentage of infants with anti-tetanus toxoid IgG concentrations ≥0.1 IU/mL
Exploratory_Non-interference | 1 month after the 2nd dose with respect to baseline titers
  Proportion of subjects with 4-fold increase in anti-pertussis IgG concentration
Exploratory_Non-interference | 1 month after the 2nd dose.
  Percentage of infants with anti Haemophilus influenzae type b (PRP) IgG concentration ≥0.15 µg/mL
Exploratory_Non-interference | 1 month after the 2nd dose.
  Percentage of infants with anti Hepatitis B surface antigen (hBsAg) IgG oncentrations ≥10 mIU/mL
Exploratory_Non-interference | 1 month after the 2nd dose.
  Percentage of infants with anti poliovirus types 1, 2 and 3 neutralizing antibody titers ≥1:8 measured

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - RSUP Prof. Dr. I.G.N.G Ngoerah, Denpasar, Bali
  - Ilmu Kesehatan anak FKUI RSCM, Jakarta Pusat, Jakarta Special Capital Region

IPD SHARING:
Plan to Share IPD: No